CLINICAL TRIAL: NCT00389532
Title: Annual Study for Serum Collection and Evaluation of Safety and Immunogenicity of Fluzone® Influenza Virus Vaccine (2006-2007 Formulation)
Brief Title: Phase IV Trial to Determine the Safety and Immunogenicity of the WHO Formulation of the 2006-2007 Fluzone® Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC35
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2009-03-30 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza; Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): aged 19 to 59 years
  Interventions: Biological: Influenza Virus Vaccine (2006-2007 Fluzone® vaccine)
- 2 (Experimental): aged ≥ 60 years
  Interventions: Biological: Influenza Virus Vaccine (2006-2007 Fluzone® vaccine)

INTERVENTIONS:
Biological: Influenza Virus Vaccine (2006-2007 Fluzone® vaccine) — Influenza vaccine
  Other Names: 2006-2007 Fluzone® vaccine
  Arms: 1
Biological: Influenza Virus Vaccine (2006-2007 Fluzone® vaccine) — Influenza vaccine
  Other Names: 2006-2007 Fluzone® vaccine
  Arms: 2

SUMMARY:
To submit remaining available sera to Center for Biologics Evaluation and Research (CBER) for further analysis by the Food and Drug Administration (FDA), the Center for Disease Control and Prevention (CDC) and the World Health Organization (WHO) to support selection and recommendation of antigen strains for subsequent influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 18 years or older on the day of inclusion.
* Participant able to attend scheduled visits and to comply with the study procedures during the entire duration of the study.
* Participant is in reasonably good health as assessed by the investigator.
* Participant willing and able to meet protocol requirements.
* Participant willing and able to give informed consent.
* For a woman, inability to bear a child or negative serum/urine pregnancy test.

Exclusion Criteria:

* Self-reported allergy to egg proteins, chicken proteins, or one of the constituents of the vaccine, such as thimerosal or formaldehyde.
* An acute illness with or without fever (temperature ≥ 99.5 °F oral) in the 72 hours preceding enrollment in the trial.
* Clinically significant findings in vital signs (including temperature ≥ 99.5 °F oral) on review of systems.
* Self-reported history of severe adverse event to any influenza vaccine.
* Laboratory-confirmed influenza infection or vaccination against influenza in the 6 months preceding enrollment in the study.
* Any vaccination in the 14 days preceding enrollment in the study or scheduled between Visit 1 and Visit 3.
* Vaccination planned in the 4 weeks following Fluzone® vaccination at Visit 1.
* Participation in any other interventional drug or vaccine trial within the 30 days preceding or during enrollment into this study.
* Immunocompromising or immunosuppressive therapy (including systemic steroid use for 2 weeks or more), cancer chemotherapy, or radiation therapy at the time of enrollment, planned during the period of this study, or at any time within the past 6 months.
* Receipt of blood or blood products within the 3 months preceding enrollment in the study.
* Diabetes mellitus requiring pharmacological control.
* Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine.
* Person deprived of freedom by an administrative or court order (having legal or medical guardian).
* For women of childbearing potential, a positive urine pregnancy test, breast feeding, or not using a medically approved form of contraception for the duration of the trial.
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Prior personal history of Guillain-Barré syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from October through December 2006 in 1 medical clinic in the US
Pre-assignment Details: A total of 116 participants that met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Aged 18 to 59 Years: Participants aged 18 to 59 years at enrollment
- Aged ≥ 60 Years: Participants aged 60 years and older at enrollment
Period: Overall Study
Arm/Group | Aged 18 to 59 Years | Aged ≥ 60 Years
Started | 60 | 56
Completed | 60 (3 of the participants did not have valid post-vaccination serological results) | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aged 18 to 59 Years | Aged ≥ 60 Years | Total
Number analyzed (Participants) | 60 | 56 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 9 | 69
  >=65 years | 0 | 47 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (12.25) | 76.4 (8.55) | 57.3 (21.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 37 | 86
  Male | 11 | 19 | 30
Region of Enrollment [Number; unit: participants]
  United States | 60 | 56 | 116

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection Site or Systemic Reaction(s) After Fluzone® Vaccination
Description: Percentage of Participants with Solicited Injection Site or Systemic Reaction(s) within 0-3 days after vaccination with Fluzone® (2006-2007 formulation)
Time Frame: 0-3 days post-vaccination
Population: Analysis was on all enrolled and vaccinated participants, Intend-to-treat population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aged 18 to 59 Years | Aged ≥ 60 Years
Number analyzed (Participants) | 60 | 56
Percentage of Participants
  Any Solicited Injection Site Reaction | 78 | 38
  Any Pain | 78 | 30
  Grade 3 Pain (Incapacitating) | 0 | 0
  Any Redness | 7 | 9
  Grade 3 Redness (≥ 5.0 cm) | 0 | 4
  Any Swelling | 3 | 6
  Grade 3 Swelling (≥ 5.0 cm) | 0 | 0
  Any Solicited Systemic Reaction | 49 | 29
  Any Fever | 3 | 2
  Grade 3 Fever (> 102.2°F) | 0 | 0
  Any Headache | 39 | 11
  Grade 3 Headache (Prevented daily activities) | 2 | 0
  Any Malaise | 25 | 9
  Grade 3 Malaise (Prevented daily activities) | 2 | 0
  Any Myalgia | 27 | 21
  Grade 3 Myalgia (Prevented daily activities) | 2 | 0

2. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition Antibodies Pre-vaccination and Post-vaccination
Description: GMTs and their 95% confidence intervals for each of the 3 antigens in the Fluzone® vaccine (2006-2007 formulation) pre-vaccination and 21 days post-vaccination.
Time Frame: 21 days post-vaccination
Population: Geometric Mean Titers were evaluated in the per-protocol immunogenicity Population
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Aged 18 to 59 Years | Aged ≥ 60 Years
Number analyzed (Participants) | 55 | 55
Titer
  H1N1 FLU A/NEW CALEDONIA/20/99 - PRE | 66.2 [41.6 to 105] | 36.9 [28.5 to 47.7]
  H1N1 FLU A/NEW CALEDONIA/20/99 - POST | 214 [151 to 304] | 77.0 [57.9 to 102]
  H3N2 FLU A/WISCONSIN/67/2005 - PRE | 67.9 [44.4 to 104] | 110 [70.8 to 170]
  H3N2 FLU A/WISCONSIN/67/2005 - POST | 453 [334 to 613] | 513 [363 to 726]
  B FLU B/MALAYSIA SPLIT/2506/2004 - PRE | 117 [83.5 to 165] | 195 [157 to 241]
  B FLU B/MALAYSIA SPLIT/2506/2004 - POST | 788 [589 to 1054] | 597 [477 to 748]

ADVERSE EVENTS:
Time Frame: Up to 28 days post-vaccination
Arm/Group | Aged 18 to 59 Years | Aged ≥ 60 Years
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/56
Other Adverse Events (participants affected / at risk) | 15/60 | 2/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aged 18 to 59 Years (N=60) | Aged ≥ 60 Years (N=56)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Headache (Nervous system disorders) | 7 (9) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.